CLINICAL TRIAL: NCT02846168
Title: The Association of Plasma Levels of GLP1 With Prognosis of Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Brief Title: Plasma GLP1 and Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Jing Wei, MD, Dr., Chinese PLA General Hospital
Other Study IDs: GLP1-AMI
Record Dates: First submitted 2016-04-12; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Angiography; Glucagon-Like Peptide 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the predicting role of plasma GLP1 level on major adverse cardiovascular events (MACE) in patients with acute myocardial infarction who undergo percutaneous coronary intervention.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is associated with high mortality and its prognosis differed among patients. Primary percutaneous coronary intervention (pPCI) is an effective method to treat AMI. To accurately predict adverse outcomes following pPCI in patients with AMI will help doctors develop precise therapeutic strategy in advance. At present how to predict adverse events before pPCI is still controversial. In our previous studies, the investigators found that glucagon like peptide -1 (GLP-1) can improve cardiac function in patients with AMI after PCI, other studies have reported that plasma GLP-1 levels is negatively correlated with CK-MB in patients with AMI, but the relationship between plasma GLP1 and prognosis of AMI patients after PCI has not been reported, the investigators hypothesized that plasma levels of GLP1 is associated with major adverse cardiovascular events (MACE) after pPCI. The investigators planned to evaluate the predicting role of plasma GLP1 level on major adverse cardiovascular events (MACE) in patients with acute myocardial infarction who undergo percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were 18 years or older and presented within 12 h from the onset of symptoms and signs of acute myocardial infarction to the catheterization laboratory.

Exclusion Criteria:

* Taking drugs of GLP-1 analogue and DPP4 inhibitor
* Cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with AMI who were admitted to the Chinese PLA General Hospital for pPCI
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events (MACE) after 6 months | at 6 months

SECONDARY OUTCOMES:
left ventricular ejection fractions | at 3 months
  measured by transthoracic echocardiography at 3 months .

CONTACTS AND LOCATIONS:
Overall Officials: Yun Dai Chen, M.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Li Jing-Wei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen WR, Hu SY, Chen YD, Zhang Y, Qian G, Wang J, Yang JJ, Wang ZF, Tian F, Ning QX. Effects of liraglutide on left ventricular function in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. Am Heart J. 2015 Nov;170(5):845-54. doi: 10.1016/j.ahj.2015.07.014. Epub 2015 Jul 26. PMID 26542491
- [Background] Chen WR, Shen XQ, Zhang Y, Chen YD, Hu SY, Qian G, Wang J, Yang JJ, Wang ZF, Tian F. Effects of liraglutide on left ventricular function in patients with non-ST-segment elevation myocardial infarction. Endocrine. 2016 Jun;52(3):516-26. doi: 10.1007/s12020-015-0798-0. Epub 2015 Nov 16. PMID 26573925
- [Background] Chen WR, Tian F, Chen YD, Wang J, Yang JJ, Wang ZF, Da Wang J, Ning QX. Effects of liraglutide on no-reflow in patients with acute ST-segment elevation myocardial infarction. Int J Cardiol. 2016 Apr 1;208:109-14. doi: 10.1016/j.ijcard.2015.12.009. Epub 2015 Dec 15. PMID 26849684